CLINICAL TRIAL: NCT04460625
Title: Investigation of the Effect of Different Blood Groups on the Survival of Intensive Care Patients
Brief Title: Effect of Blood Group on the Survival Status of Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sibel Köstekli, Zonguldak Bülent Ecevit University Faculty of Health Sciences, Zonguldak Bulent Ecevit University
Other Study IDs: 2020-09
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Critical Illness; Nurse's Role; Risk Factor; Prognosis
Keywords: intensive care; intensive care nursing; critical patient; blood group; survival
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research was planned to determine the effect of different blood groups on the 90-day survival of intensive care patients who were treated and maintained for the first time in the intensive care unit.

The research is a retrospective descriptive research. For the first time in an intensive care unit aged 18 and over, between January 1, 2014 and December 31, 2019, of a state and a university hospital in the Western Black Sea Region, in intensive care units (both medical and surgical patients), All the patients, who were hospitalized in the intensive care unit for at least 24 hours, were discharged from the intensive care unit for 90 days and less, and all the information in the Patient Information Form can be accessed from the automation system.

The research will be conducted between 01.04.2020-01.07.2020 by collecting the necessary data within the 'Patient Information Form' of the patients from the information processing unit of the hospitals where the research will be conducted.

DETAILED DESCRIPTION:
Intensive care units; They are units where advanced technological tools and equipment are used to provide the highest level of benefit to life-threatened patients, and physicians and nurses specializing in the treatment and care of patients are involved. Intensive care patients; '' To prevent patients who are at risk due to physiological decompensation and patients who are physically physiologically fluctuating, need a treatment to be carried out with the harmony between physician and nurse to ensure survival, the application of this treatment without showing waves, especially details and care, and unexpected adverse events. and patients who require continuous monitoring to provide immediate intervention by the intensive care team. Intensive care patients, as can be understood from the definition, are the patients whose general conditions change rapidly due to the presence of a life-threatening condition, due to the impact of several systems that require close monitoring and control vital functions.

Respiratory, cardiovascular, neurological, etc. Many conditions, such as chronic diseases, genetic, individual and environmental factors, of patients who are in danger of life due to many important health problems can affect the prognosis of the patients. In addition to these factors, although there is insufficient evidence, blood groups are reported to be effective in the survival of intensive care patients. Whatever the underlying situation is, the most important thing is undoubtedly the blood for the maintenance of a healthy life. It is known to affect human health in many cases, from the amount of blood circulating in the vein to the structure of blood cells.

It was found for the first time in the years of 1899 and 1900 that human blood differs from individual to individual due to some physiological features. These different blood groups discovered are A, B and AB. Later, with the discovery of the Rh factor along with the O (zero) blood group, studies on the effects and differences of blood groups on humans have increased rapidly. Today, studies on the relationship between blood groups and diseases are ongoing.

As a result of some studies; It has been determined that the AB blood group plays a role as a risk factor in both venous thromboembolism and coronary artery disease. The risk of both arterial and venous thrombotic events in the AB blood group There is evidence that it has high levels of vonWillebrand factor (vWF) and factor VIII. Depending on the limitation of mobilization in intensive care patients, it may increase the negative effect of the blood group on the patient compared to the patients hospitalized in other clinics. However, in patient groups with a high risk of bleeding, this may provide additional benefit for patients with AB blood group with higher levels of vonWillebrand factor (vWF) and factor VIII. In their research, Franchini et al. Reported that bleeding rate increased significantly in patients with O blood group, especially in surgical procedures with high risk of blood loss. Therefore, it has been observed that patients with AB blood group are more likely to survive after major heart surgery and this situation is explained in relation to the decrease in the number of blood transfusions. The results of metaanalysis study of Dentali et al. Also pointed out that having an O blood group in terms of bleeding may be an important genetic factor. It is important that the intensive care nurse includes this information in patient care.

In a study conducted to determine the link between ABO blood group, lipid profiles and coronary artery disease and to determine the effect size of the link, patients in the A blood group were found to have higher total cholesterol rates while lower LDL rates. Jiang et al; They found that ABO blood groups were not associated with age, gender, and blood pressure in stable coronary artery patients undergoing percutaneous coronary intervention, but blood groups were associated with 2-year cardiac death.

Although it is known that genetic diversity affecting the prognosis of patients is a factor in determining survival after being taken into intensive care, it can be difficult and costly to evaluate in a short time in clinical practice. Also, to predict the prognosis of critical patients in intensive care units today. it is still very difficult. In this context, individualized medicine; It can provide a better understanding of patients' risks arising from genetic, environmental and social factors and better planning of the results of treatment. At the onset of critical illness, knowing all possible risk factors to effectively manage patients creates a chance to achieve more successful treatment and care outcomes. more difficult to determine the effect on survival of genetic diversity, although there is nothing for a long time consuming and costly, ABO blood group of the survival effect according to the risk classification system, the addition of both easier, additional benefits to the patient to be quickly and cost-free by the Ministry of Health in sağlayabilir. Türkiye APACHE II (Acute Physiology and Chronic Health Evaluation) is the most commonly used scale to calculate the expected mortality rate according to the severity of the disease that is approved and admitted to intensive care.

The relationship between patients' blood groups and mortality is thought to exist as a result of research. In the research of Slade et al; After the patients were admitted to the intensive care unit, the relationship between blood groups and mortality was evaluated in the 90-day period; It has been determined that patients with intensive care with AB blood group have a higher 90-day survival time compared to other blood group patients. In line with this result, there is a need for studies for the risk assessment scales and the addition of the blood group factor for intensive care patients.

Quality nursing care is an important factor affecting the prognosis of patients. It is predicted that the application of individualized patient care will positively affect the physiological, psychological and social health of the patient. Nurses are healthcare professionals who are in key condition next to the patient in any case in intensive care units. Higher quality care of nurses at the center of many interventions in the intensive care unit has been associated with improved patient outcomes, including mortality. In line with this information, the research was planned to determine the effect of different blood groups on the 90-day survival of intensive care patients who were treated and maintained for the first time in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or older
* Being in the intensive care unit for the first time,
* To stay in the intensive care unit for at least 24 hours.
* Being discharged from the intensive care unit in 90 days and less
* All information in the Patient Information Form can be accessed from the automation system.

Exclusion Criteria:

* Being under the age of 18
* Having previously slept in the intensive care unit
* Intensive care hospitalization has ended in less than 24 hours.
* Staying in the intensive care unit for more than 90 days
* Failure to reach all questions in the Patient Information form from the automation system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Zonguldak Atatürk State Hospital located in the Western Black Sea Region, were treated between January 1, 2014 and 31.12.2019 in intensive care units (both medical and surgical patients). The number of patients admitted to the intensive care units was determined from the information processing unit of the hospitals and determined as 4.120. These patients will form the universe of the research. Of these patients; All patients who are hospitalized for the first time in the intensive care unit, who are in the intensive care unit for at least 24 hours, who are discharged from the intensive care unit for 90 days and less, all information in the data collection form, 18 years of age and over, will be the sample group.
Sampling Method: Non-Probability Sample
Enrollment: 3114 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Examination of the correlation between blood group of patients and rh factor and secondary complication development during admission to intensive care units | Whether or not complications develop within 90 days of admission to patients in intensive care unit
  At the onset of critical illness,knowing all possible risk factors to effectively manage patients creates a chance to achieve more successful treatment and care outcomes.Although it is more difficult time consuming and costly to determine the effect of genetic diversity on survival,the addition of ABO blood groups to the risk classification system according to the effect on survival may also provide additional benefits to the patient as it will be easier,faster and inexpensive.It is observed that this factor is missing in the mortality risk diagnosis forms used during the intensive care hospitalization currently used.Patients with 0 blood group,in which the AB blood group plays a role in both venous thromboembolism and coronary artery disease as a risk factor and their tendency to clot;It has been reported that the bleeding rate increases significantly,especially in surgical procedures with high risk of blood loss.If it is considered that the procedures applied in intensive care ünit.
Examining the correlation between the patient's blood group and rh factor and mortality in patients | Mortality rates will be checked within 90 days from the patients' admission to intensive care unit.
  The relationship between patients' blood groups and mortality is thought to exist as a result of research. In a research; After the patients were admitted to the intensive care unit, the relationship between blood groups and mortality was evaluated in the 90-day period; It has been determined that patients with intensive care with AB blood group have a higher 90-day survival time compared to other blood group patients. In line with this result, there is a need for studies for the risk assessment scales and the addition of the blood group factor for intensive care patients.

SECONDARY OUTCOMES:
Examination of the correlation between patients 'invasive mechanical ventilation status and duration, and patients' 90-day survival | 90 days
  Patients receiving invasive mechanical ventilator support is a risk factor for morbidity and mortality. Because, patients who receive mechanical ventilation support increase the risk of complications compared to other patients. In the research, the status and duration of patients receiving mechanical ventilator support will be recorded with the patient information form and it is planned to look at the relationship between the appropriate statistical methods at the end of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Köstekli, Principal Investigator — Zonguldak Bülent Ecevit University Faculty of Health Sciences Nursing Department
Locations (1):
- Zonguldak Atatürk State Hospital, Zonguldak, Meşrutiyet, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No